CLINICAL TRIAL: NCT01830439
Title: A Phase 1, Randomized, Balanced, Single-Dose, Two-Period, Two-Sequence, Crossover, Open-Label Study of the Effect of Food on the Bioavailability and Pharmacokinetics of PA-824 Tablets in Healthy Adult Subjects
Brief Title: Food Effect Study on the Bioavailability and PK of PA-824 Tablets in Healthy Adult Subjects (CL-009)
Acronym: CL-009
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PA-824-CL-009
Record Dates: First submitted 2013-02-12; First posted 2013-04-12 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Tuberculosis
Keywords: tuberculosis; PK; PA-824; food effect; pretomanid; CL-009
MeSH Terms: conditions — Tuberculosis | interventions — pretomanid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fed PA-824 200mg (Experimental): 200 mg PA-824 (4 x 50 mg tablets) in Phase A was administered 30 minutes after the start of a high-calorie, high-fat breakfast provided after a minimum 10-hour overnight fast and was administered with 240 mL tap water.
  Interventions: Drug: PA-824 200mg
- Fasted PA-824 200 mg (Experimental): 200 mg PA-824 (4 x 50 mg tablets) in Phase A was administered 30 minutes after a minimum 10-hour overnight fast and was administered with 240 mL tap water.
  Interventions: Drug: PA-824 200mg
- Fed PA-824 50mg (Experimental): 50 mg PA-824 (1 x 50 mg tablets) in Phase B was administered 30 minutes after the start of a high-calorie, high-fat breakfast provided after a minimum 10-hour overnight fast and was administered with 240 mL tap water.
  Interventions: Drug: PA-824 50mg
- Fasted PA-824 50mg (Experimental): 50 mg PA-824 (1 x 50 mg tablets) in Phase B was administered after a minimum 10-hour overnight fast and was administered with 240 mL tap water.
  Interventions: Drug: PA-824 50mg

INTERVENTIONS:
Drug: PA-824 200mg — Two single administrations of 200mg PA-824 each administered by four 50mg tablets, one administered in the fed state and one administered in the fasted state. The two administrations were separated by 8 days.
  Arms: Fasted PA-824 200 mg; Fed PA-824 200mg
Drug: PA-824 50mg — Two single administrations of 50mg PA-824 each administered by one 50mg tablet, one administered in the fed state and one administered in the fasted state. The two administrations were separated by 8 days.
  Arms: Fasted PA-824 50mg; Fed PA-824 50mg

SUMMARY:
This will be a Phase 1, single-center, randomized, balanced, single-dose, two-period, two-sequence, crossover, open-label study to evaluate the effect of food on the pharmacokinetics of PA-824. The hypothesis to be tested in this study is that the rate and extent of absorption of two doses of PA-824 (50mg or 400 mg and 200mg) are the same after a high-calorie, high-fat meal as compared with after a minimum 10-hour fast.

For each of the two dose levels 16 subjects with approximately 8 men and 8 women, will be enrolled for a total of 32 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, have provided written informed consent (as evidenced by signature on an informed consent document approved by an IRB), and agree to abide by the study restrictions.
2. Be healthy non-tobacco/nicotine using (6-month minimum) adult subjects, 19 to 50 years of age, inclusive.
3. Be medically healthy subjects with clinically insignificant Screening results (among laboratory profiles, medical histories, ECGs, or physical exam), as deemed by the Principal Investigator.
4. Have a body mass index of 18 to 29.
5. Have negative urine test results for alcohol and drugs of abuse such as amphetamines, cannabinoids, and cocaine metabolites at both Screening and Check-in.
6. Agree to follow the requirements set forth in the protocol regarding pregnancy controls and donation of sperm, blood, or blood components.

Exclusion Criteria:

1. Any clinically significant (as deemed by the Principal Investigator) history, acute illness (resolved within 4 weeks of screening), or presence of cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal (including eating disorders), endocrine, metabolic, immunologic, dermatologic, neurologic, psychological, or psychiatric disease.
2. History of peptic ulcer disease, gastritis, esophagitis, or gastroesophageal reflux disease.
3. History of any cardiac abnormality (as deemed by the Principal Investigator).
4. Any clinically significant ECG abnormality at Screening (as deemed by the Principal Investigator and the Sponsor's Medical Monitor). Note: the following can be considered not clinically significant without consulting Sponsor's Medical Monitor:

   * Sinus bradycardia with heart rate ≥50 beats per minute (sinus bradycardia with heart rate between 45 and 49, inclusive, is acceptable only in younger athletic subjects)
   * Mild first degree A-V block (P-R interval <0.23 sec)
   * Right or left axis deviation
   * Incomplete right bundle branch block
   * Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic subjects
5. History of prolonged QT interval.
6. Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease or CHF or terminal cancer)
7. Resting pulse rate < 40 or > 100 bpm at Screening.
8. At Screening blood pressure greater than 140/90 mm Hg or below 95/65 mm Hg (supine, after a minimum 5-minute supine rest)
9. At either Screening or the pre-dose read before the first dose, a QTcB (Bazett's correction) >450ms for men and women, calculated from the average of triplicate reads collected at one sitting.
10. At either Screening or the pre-dose read before the first dose, a QTcF (Fridericia's correction) >450ms for men and women, calculated from the average of triplicate reads collected at one sitting.
11. History of hypokalemia or hypomagnesemia.
12. History or presence of alcoholism or drug abuse within the past 2 years (as deemed by the Principal Investigator).
13. Use of alcohol within 72 hours prior to dosing.
14. Significant history of drug and/or food allergies (as deemed by the Principal Investigator).
15. For women, subject is pregnant (positive test for serum HCG at Screening or Check-in), breastfeeding or planning to conceive a child within 1 week of cessation of treatment.
16. For males, planning to father a child within 12 weeks of cessation of treatment.
17. History of lens opacity or evidence of lens opacity on slit lamp ophthalmologic examination.
18. Any contraindication to the use of nitroimidazoles or prior treatment with PA-824 or OPC-67683.
19. Use of any systemic or topical prescription medication within 14 days prior to dosing or during the study, except hormonal contraceptives in women
20. Use of any systemic or over-the-counter medication including vitamins, herbal preparations, antacids, cough and cold remedies, etc., within 7 days prior to dosing or during the study.
21. Use of any drugs or substances within 30 days prior to dosing known to be strong inhibitors or inducers of cytochrome P450 enzymes (including quinidine, tyramine, ketoconazole, testosterone, quinine, gestodene, metyrapone, phenelzine, doxorubicin, troleandomycin, cyclobenzaprine, erythromycin, cocaine, furafylline, cimetidine, dextromethorphan, etc.) or known to prolong the QT interval (including amiodarone, bepridil chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, quinolones, sotalol, sparfloxacin, thioridazine,) or barbiturates, opiates, or phenothiazines.
22. Use of any therapeutic agents known to alter any major organ function (e.g., barbiturates, opiates, phenothiazines, cimetidine, etc.) within 30 days prior to dosing.
23. Consumption of products containing grapefruit within 10 days prior to dosing.
24. Any special dietary changes during the 30 days prior to dosing, as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor.
25. Any strenuous exercise within 7 days of Check-in, as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor.
26. Donation of whole blood or significant loss of blood within 56 days prior to dosing.
27. Plasma donation within 7 days prior to dosing
28. Participation in another interventional clinical trial within 30 days prior to dosing.
29. Any serum creatinine or BUN measure beyond the upper limit of the normal range at Screening or Check-in. Individual values may be discussed with the Sponsor Medical Monitor.
30. Hemoglobin < 12.0 g/dL at the screening and check-in visit.
31. Positive Screening test for HCV, HBV, or HIV.
32. Any other factor which suggests to the Principal Investigator that the subject should not participate in the study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Time of the maximum drug concentration in hours [Tmax] | mean through 36 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours post dose
  To compare the rate and extent of absorption as measured by Tmax of a single oral dose of PA-824 tablets (200 mg in Phase A and either 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. Tmax is obtained without interpolation.
Maximum observed drug concentration in ng/mL [Cmax] | mean through 36 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours post dose
  To compare the rate and extent of absorption as measured by Cmax of a single oral dose of PA-824 tablets (200 mg in Phase A and either 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast.
Area under the drug concentration-time curve in ng*hr/mL [AUC(0-t)] | mean through 36 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours post dose
  To compare the rate and extent of absorption as measured by AUC(0-t) of a single oral dose of PA-824 tablets (200 mg in Phase A and either 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. AUC(0-t) is calculated using linear trapezoidal summation from time zero to time t, where t is the time of the last measurable concentration.
Area under the drug concentration-time curve from time zero to infinity in ng*hr/mL [AUC(0-inf)] | mean through 36 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours post dose
  To compare the rate and extent of absorption as measured by AUC(0-inf) of a single oral dose of PA-824 tablets (200 mg in Phase A and either 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. AUC(0-inf) is calculated as AUC(0-t) + Ct/Kel.

SECONDARY OUTCOMES:
Ratio of AUC(0-t) to AUC(0-inf) [AUC(0-t)/ AUC(0-inf)] | mean through 36 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours post dose
  To compare AUC(0-t)/ AUC(0-inf) of a single oral dose of PA-824 tablets (200 mg in Phase A and 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast.
Number of participants with adverse events | through the study Day 13, and through Day 103 for SAE and ophthalmologic events
  To compare the safety and tolerability as measured by the number of participants with adverse events after a single oral dose of PA-824 tablets (200 mg in Phase A and 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast.
Elimination half-life in hours [t1/2] | mean through 36 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours post dose
  To compare t1/2 of a single oral dose of PA-824 tablets (200 mg in Phase A and 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. T1/2 is calculated as ln (2)/Kel.
Terminal elimination rate constant in 1/hour [Kel] | mean through 36 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours post dose
  To compare Kel of a single oral dose of PA-824 tablets (200 mg in Phase A and 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. Kel is calculated by linear regression of the terminal linear portion of the log concentration vs. time curve, using at least 3 data points
Oral clearance in L/hour [Cl/F] | mean through 36 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours post dose
  To compare Cl/F of a single oral dose of PA-824 tablets (200 mg in Phase A and 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. Cl/F is calculated as Dose/AUC(0-inf).
Volume of distribution following oral administration in L [Vd/F] | mean through 36 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours post dose
  To compare Vd/F of a single oral dose of PA-824 tablets (200 mg in Phase A and 50 mg or 400 mg in Phase B) in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. Vd/F is calculated as (CL/F)/Kel.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — MDS Pharma Services (Celerion)
Locations (1):
- MDS Pharma Services (Celerion), Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Winter H, Ginsberg A, Egizi E, Erondu N, Whitney K, Pauli E, Everitt D. Effect of a high-calorie, high-fat meal on the bioavailability and pharmacokinetics of PA-824 in healthy adult subjects. Antimicrob Agents Chemother. 2013 Nov;57(11):5516-20. doi: 10.1128/AAC.00798-13. Epub 2013 Aug 26. PMID 23979737
- See also: Global Alliance for TB Drug Development website — http://www.tballiance.org